CLINICAL TRIAL: NCT05284708
Title: The "USAbility" Study - Human Factor Validation Testing of the Atalante Exoskeleton
Brief Title: Atalante USAbility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wandercraft (Industry)
Collaborators: Innovative Medical Technologies, Inc (Other); Shirley Ryan AbilityLab (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP003
Record Dates: First submitted 2021-11-23; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Hemiplegia
Keywords: Exoskeleton
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Intervention Model Description: Single Group Usability Observational Study, Operators
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Clinical Operators (Other): Experimental: 15 healthcare professionals will be recruited for the study. The group includes physiotherapists (PTs), physiotherapist assistants (PTAs), clinical exercise physiologists (EPs), and rehabilitation technicians (RTs), all resident in US and representing the final users of the device. Operators are representative of the final users of the exoskeleton.
  Interventions: Device: Atalante

INTERVENTIONS:
Device: Atalante — Powered Exoskeleton

SUMMARY:
The "USAbility" study - Human Factor Validation Testing of the Atalante exoskeleton aims at demonstrating that Atalante can be used by the intended users without serious use errors or problems, for the intended uses and under the expected use conditions.

DETAILED DESCRIPTION:
Robotic assisted rehabilitation has been successfully proposed and employed especially when motor conditions do not allow the patient to walk. However, limitations in usability often prevent from a widespread adoption of robotic devices (e.g., exoskeletons) in clinical routine Their success is highly dependent on user acceptance, which in turn is determined by the subjective intention-to-use, as well as by the perception of usability and comfort. Approaching the design of such devices with Human Factors and Usability engineering has proven to be an effective means to enhance performance-related outcomes such as fewer errors, less time and lower mental effort. Usability testing is commonly considered a cornerstone in user-centered design, as it provides information about problematic design issues. It further serves as a validation test for performance requirements, such as efficiency or safety of operation.

Based on these considerations, we propose a study to analyze the usability of Atalante device and demonstrate that it can be used by the intended users without serious use errors or problems, for the intended uses and under the expected use conditions. The scope of this research study is to validate all the critical tasks performed by the intended operators of the device in a typical rehabilitation session according to IEC 62366-1(2020) and the FDA Guidance "Applying human Factors and Usability Engineering to Medical Devices". This knowledge will inform further development of exoskeletons and improve the widespread uptake and medical use of such devices, in light of the many benefits that these technologies can bring to future patients.

15 operators will be recruited and attend an 8 hours and 30 minutes training split in three days and provided by Wandercraft before the use of the device.

Usability will be assessed by:

1. IFU questionnaire
2. Simulated tasks test: users' performance will be observed to determine if the assigned task was performed correctly by the operator. 5 patients will be recruited to simulate a typical session with the exoskeleton*.
3. Final debriefing: subjective operators' assessments will be collected after the test The device user interfaces represent the final design of the device, and the study will be performed in actual conditions of use at the Shirley Ryan Ability Lab, a physical medicine and rehabilitation research hospital based in Chicago, Illinois, USA which is representative of the intended use environment.

   * Patients performance is out of the scope of the evaluation

ELIGIBILITY:
Inclusion Criteria:

Operators*

* Operators belonging to one of the following categories:

  * Physiotherapists
  * Physiotherapist assistants
  * Exercise physiologists
  * Rehabilitation technicians
* Operators are US residents
* Operators can speak, write, and understand English

  * Need for supervision for specific operators' categories is regulated by the specific state laws and jurisdiction and is part of the responsibility of the healthcare facility.

Patients:

* Aged 18 and over
* More than 30 days post stroke
* English speakers: able to read, understand, and sign the informed consent
* With specific morphological characteristics

Exclusion Criteria:

Patients:

* Individuals with severe spasticity of adductor muscles, hamstring, quadriceps, and triceps surrae. Severe spasticity is defined by a score greater than 3 on the modified Ashworth scale
* Pregnant women
* History(ies) of osteoporotic fracture(s) and/or treatment causing secondary osteoporosis
* Pressure Ulcer of Grade I or higher according to the NPUAP International Pressure Ulcer Classification System - EPUAP, in areas of contact with the Atalante system
* Cognitive impairment that prevents the patient from understanding instructions, at the physician's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Observational Usability - Critical Tasks | 10.5 hours
  The primary usability objective that will serve as acceptance criterion for this test is 100% of recruited operators complete each of the critical tasks successfully.

SECONDARY OUTCOMES:
Observational Usability - Non-Critical Tasks and IFU and training assessment | 10.5 hours
  Secondary Outcome Measures include 90% of recruited operators can respond to the IFU questionnaire correctly and is considered "passed" if the operator can correctly answer 9 out 10 questions in the provided time and 90% of recruited operators can complete each of the non-critical tasks successfully and 90% of recruited operators rates the training and associated documents as 3 or higher on a 5-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: M4 Study — https://clinicaltrials.gov/ct2/show/NCT04110561?term=atalante+exoskeleton&draw=2&rank=3
- See also: SPIRIT Study — https://clinicaltrials.gov/ct2/show/NCT04187209?term=atalante+exoskeleton&draw=2&rank=2
- See also: INSPIRE Study — https://clinicaltrials.gov/ct2/show/NCT04694001?term=atalante+exoskeleton&draw=2&rank=1